CLINICAL TRIAL: NCT06903000
Title: Effects of Instrument-Assisted Soft Tissue Mobilization and Vibration Therapy on Pain, Functional Status, Proprioception, and Kinesiophobia in Individuals With Cervical Disc Herniation
Brief Title: Effects of IASTM and Vibration Therapy in Cervical Disc Herniation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emre DANSUK (Other)
Responsible Party: Sponsor-Investigator, Emre DANSUK, Principal Investigator, Medipol University
Organization: Medipol University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E-10840098-202.3.02-1924
Record Dates: First submitted 2025-03-24; First posted 2025-03-30 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Intervertebral Disc Displacement; Neck Pain
Keywords: Cervical disc herniation; Neck pain; Instrument-assisted soft tissue mobilization; Vibration therapy; Proprioception; Kinesiophobia; Physiotherapy
MeSH Terms: conditions — Intervertebral Disc Displacement; Neck Pain; Kinesiophobia

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Vibration Therapy Group (Experimental): Participants in this group will receive percussion-based vibration therapy applied using a percussion massage device (Compex Fix 2.0) with a soft head attachment. Therapy will target trapezius, levator scapula, and cervical paravertebral muscles along their origin-insertion lines for 3 minutes per muscle group. Sessions will be conducted 3 days per week over 3 weeks, alongside conventional physiotherapy, including heat therapy (20 min), Transcutaneous Electrical Nerve Stimulation (TENS - 100 Hz), range-of-motion (ROM) exercises (2 sets of 10 repetitions, 2-second holds at end-range), and isometric strengthening exercises (2 sets of 10 repetitions, 6-second holds per direction).
  Interventions: Device: a percussion massage gun; Other: Conventional Exercise Group (Control)
- Instrument-Assisted Soft Tissue Mobilization (IASTM) Group (Experimental): Participants will receive instrument-assisted soft tissue mobilization applied using specially designed stainless-steel instruments. Techniques (Sweep, Fan, Brush) will be applied to cervical and upper-back musculature (splenius, suboccipital, upper-middle-lower trapezius) and related fascia between C1-T1 vertebrae, parallel to muscle fibers for approximately 6 minutes per session. Each technique will consist of 8-10 repetitions. Treatments will occur 3 sessions per week for 3 weeks, alongside conventional physiotherapy interventions (heat therapy for 20 minutes, TENS at 100 Hz, ROM exercises, and isometric strengthening exercises as described above).
  Interventions: Device: specially designed stainless-steel instruments; Other: Conventional Exercise Group (Control)
- Conventional Exercise Group (Control) (Active Comparator): Participants in this control group will receive conventional physiotherapy treatment alone. The treatment includes heat therapy applied to the cervical region for 20 minutes, TENS application at a frequency of 100 Hz to painful areas, ROM exercises performed in all cervical directions (2 sets of 10 repetitions, 2-second holds at end-range), and isometric strengthening exercises in cervical flexion, extension, and lateral flexion directions (2 sets of 10 repetitions, 6-second holds per repetition). Sessions will take place 4 days per week for 3 weeks.
  Interventions: Other: Conventional Exercise Group (Control)

INTERVENTIONS:
Device: a percussion massage gun — Participants in this group will receive percussion-based vibration therapy applied using a percussion massage device (Compex Fix 2.0) with a soft head attachment. Therapy will target trapezius, levator scapula, and cervical paravertebral muscles along their origin-insertion lines for 3 minutes per muscle group.
  Arms: Vibration Therapy Group
Device: specially designed stainless-steel instruments — Participants will receive instrument-assisted soft tissue mobilization applied using specially designed stainless-steel instruments. Techniques (Sweep, Fan, Brush) will be applied to cervical and upper-back musculature (splenius, suboccipital, upper-middle-lower trapezius) and related fascia between C1-T1 vertebrae, parallel to muscle fibers for approximately 6 minutes per session. Each technique will consist of 8-10 repetitions.
  Arms: Instrument-Assisted Soft Tissue Mobilization (IASTM) Group
Other: Conventional Exercise Group (Control) — Participants in this control group will receive conventional physiotherapy treatment alone. The treatment includes heat therapy applied to the cervical region for 20 minutes, TENS application at a frequency of 100 Hz to painful areas, ROM exercises performed in all cervical directions (2 sets of 10 repetitions, 2-second holds at end-range), and isometric strengthening exercises in cervical flexion, extension, and lateral flexion directions (2 sets of 10 repetitions, 6-second holds per repetition). Sessions will take place 4 days per week for 3 weeks.

SUMMARY:
This study investigates the effects of instrument-assisted soft tissue mobilization (IASTM) and percussion massage therapy on pain, functional status, proprioception, and kinesiophobia in individuals with cervical disc herniation. A total of 66 participants diagnosed with cervical disc herniation will be randomly divided into three groups: vibration therapy, IASTM, and conventional exercise. Each group will receive conventional physiotherapy, while the intervention groups will additionally receive their respective therapies. Outcomes will be measured using the Visual Analog Scale (VAS), Neck Disability Index (NDI), Laser Pointer Joint Position Sense Test, and Tampa Scale for Kinesiophobia (TSK). The aim is to evaluate and compare the effectiveness of both therapies in reducing pain, improving functionality and proprioception, and decreasing fear of movement.

DETAILED DESCRIPTION:
Cervical disc herniation is a common musculoskeletal condition that causes significant pain and functional limitations, often affecting individuals in their middle ages and those working in sedentary occupations. This study aims to investigate the therapeutic effects of two modern physical therapy techniques-Instrument-Assisted Soft Tissue Mobilization (IASTM) and percussion-based vibration therapy-on pain, functional capacity, proprioception, and kinesiophobia in individuals with cervical disc herniation.

A total of 66 participants diagnosed with cervical disc herniation will be recruited and randomly assigned to one of three groups: (1) Vibration Therapy Group, (2) IASTM Group, and (3) Conventional Exercise Group. All participants will receive standard physiotherapy, including thermotherapy, TENS, and range of motion exercises. Intervention groups will additionally receive either percussion massage therapy (3 sessions/week for 3 weeks) or IASTM (3 sessions/week for 3 weeks), targeting the cervical and upper back musculature.

Outcome measures will include the Visual Analog Scale (VAS) for pain, the Neck Disability Index (NDI) for functional assessment, a Laser Pointer Joint Position Sense Test for proprioception, and the Tampa Scale for Kinesiophobia (TSK) to assess fear of movement. The study seeks to compare the effectiveness of these approaches in improving clinical outcomes and contributing to evidence-based rehabilitation strategies for individuals with cervical disc pathology.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of cervical disc herniation.
* Have a complaint of neck pain lasting at least 3 weeks.
* Have a restriction in cervical range of motion.

Exclusion Criteria:

* Have any additional orthopedic or neurological disorders besides cervical problems.
* Have a history of previous trauma to the cervical region.
* Have received physiotherapy within the past 6 months.
* Are unable to tolerate vibration therapy.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 57 (Actual)
Dates: Start 2025-03-28 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Assessment of Joint Position Sense (Proprioception) | 3 weeks
  This assessment measures joint position sense-a component of proprioception-which provides information regarding the speed and direction of active and passive movements without visual cues.Participants will be seated at a distance of 100 cm from a target board measuring 90x80 cm. A laser pointer will be secured to the participant's head using a suitable headband. Participants will initially align the laser pointer vertically onto the center (origin) of the target board with their eyes open. They will then flex their head forward and subsequently return to the neutral position, realigning the pointer to the center. Next, participants will repeat the same process with their eyes closed. After performing cervical flexion, they will attempt to return their head to the perceived neutral position without visual assistance. The deviation from the origin will be measured and recorded as an indicator of joint position sense accuracy.

SECONDARY OUTCOMES:
Pain Assessment (Visual Analog Scale - VAS) | 3 weeks
  The Visual Analog Scale (VAS) will be used to evaluate participants' pain intensity. The VAS consists of a horizontal line measuring 10 cm, where '0' represents "no pain" and '10' represents "unbearable pain." Participants will be asked to mark the point that represents their perceived level of pain on this scale. The distance from the starting point (0 cm) to the participant's mark will be measured with a ruler and recorded.
Neck Disability Index (NDI) | 3 weeks
  The Neck Disability Index (NDI) will be used to assess participants' functional limitations related to neck pain. Developed by Vernon and Mior, the NDI is a reliable, valid, and easy-to-administer questionnaire adapted and validated for use in Turkey. It comprises 10 sections evaluating the severity of pain, lifting, reading, headaches, personal care, work activities, concentration, sleep, recreational activities, and driving. Each section offers six responses scored from 0 to 5. A score of 0 indicates no pain or functional limitation, whereas a score of 5 indicates maximum pain and severe limitation in daily activities.
Kinesiophobia Assessment (Tampa Scale for Kinesiophobia -TSK) | 3 weeks
  Participants' kinesiophobia will be assessed using the Tampa Scale for Kinesiophobia (TSK). This scale, originally developed by Kori et al. in 1990 and validated for use in Turkish, consists of 17 questions designed to measure participants' fear of movement. Responses are scored on a 4-point Likert scale: "strongly disagree" (1), "disagree" (2), "agree" (3), and "strongly agree" (4). Items 4, 8, 12, and 16 are reverse-scored before calculating the total score. Total scores range between 17 and 68, with higher scores indicating a greater degree of kinesiophobia.

CONTACTS AND LOCATIONS:
Overall Officials: Emre Dansuk, PhD, Principal Investigator — Medipol University
Locations (1):
- Emre Dansuk, Istanbul, Beykoz, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Menek B, Dansuk E, Gorguluer S. Instrument-assisted soft tissue mobilization and percussion massage therapy in cervical disc herniation: a randomized controlled study. J Orthop Surg Res. 2025 Aug 30;20(1):801. doi: 10.1186/s13018-025-06238-5. PMID 40886005